CLINICAL TRIAL: NCT06101576
Title: Readmission Following Endourological Prostatic Surgery for Benign Prostatic Obstruction: Review of 20 Years of Experience
Brief Title: Readmission Following Prostatic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: 2436
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: BPH With Urinary Obstruction
Keywords: BPH; TURP; Laser prostatectomy; BNC; Holmium Laser
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Transurethral incision of the prostate (TUIP): Patients who underwent TUIP using electrocautery or Laser.
  Interventions: Procedure: TUIP
- Transurethral resection of the prostate (TURP): Patients who underwent TURP using monopolar or bipolar electrocautery.
  Interventions: Procedure: TURP
- Prostate Vaporization: Patient who underwent vaporization of the prostate using plasma or laser energy (GreenLight PVP and Thulium vaporization of the prostate).
  Interventions: Procedure: Prostate Vaporization
- Anatomical endoscopic enucleation of the prostate (AEEP): Patient who underwent anatomical endoscopic enucleation of the prostate (AEEP) using Holmium, Thulium or GreenLight laser or bipolar current.
  Interventions: Procedure: AEEP

INTERVENTIONS:
Procedure: TUIP — Patient who underwent transurethral incision of the prostate (TUIP) using electrical current or laser beam.
  Groups: Transurethral incision of the prostate (TUIP)
Procedure: TURP — Patient who underwent transurethral resection of the prostate (TURP) using momopolar or bipolar current.
  Groups: Transurethral resection of the prostate (TURP)
Procedure: Prostate Vaporization — Patient who underwent vaporization of the prostate using plasma or laser energy (GreenLight PVP and Thulium vaporization of the prostate).
  Groups: Prostate Vaporization
Procedure: AEEP — Patient who underwent anatomical endoscopic enucleation of the prostate (AEEP) using Holmium, Thulium or GreenLight laser or bipolar current.
  Groups: Anatomical endoscopic enucleation of the prostate (AEEP)

SUMMARY:
This study will be conducted to estimate readmission rate and reasons for readmission after all modalities of endoscopic transurethral surgeries for treatment of BOO secondary to BPH in the last 20 years.

DETAILED DESCRIPTION:
Computerized patient information system (PIS) of Urology and Nephrology Center (UNC) and database of prostate unit of UNC will be reviewed for all preoperative, intraoperative and post discharge data. All follow up visits will be traced for outcome measurement. Patients with no hospital follow up visit will be contacted by phone and interrogated about their LUTS control state, ongoing medication and history of secondary procedures.

ELIGIBILITY:
Inclusion Criteria:

Men who underwent transurethral prostatic surgery for BPH causing BOO at Urology and Nephrology Center, Mansoura University, Egypt from Jun. 2005 to Dec. 2024.

Exclusion Criteria:

1. Patients who underwent TUR tunnelling for prostatic adenocarcinoma.
2. LUTS secondary to neuropathic bladder.
3. Incidentally diagnosed prostate cancer after surgery

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Study Population: They will be the subdivided into four groups:
  Group I: Patient who underwent transurethral incision of the prostate (TUIP) using electrical current or laser beam. Group II: Patient who underwent transurethral resection of the prostate (TURP) using momopolar or bipolar current. Group III: Patient who underwent vaporization of the prostate using plasma or laser energy (GreenLight PVP and Thulium vaporization of the prostate). Group IV: Patient who underwent anatomical endoscopic enucleation of the prostate (AEEP) using Holmium, Thulium or GreenLight laser or bipolar current.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The need for post discharge hospital readmission. | 90 days
  The need for post discharge hospital readmission after surgery.

SECONDARY OUTCOMES:
Differences of readmission rates | 90 days
  Difference of readmission rates for different modalities of transuretheral prostatic surgery.
Change in the causes of readmission over time. | 20 years
  Change in the causes of readmission over time.
Causes and predictors of readmission. | 90 days
  Causes and predictors of readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R EL-Nahas, MD, Principal Investigator — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No